A Phase 2a Randomised, Double Blind, Multi-centre Study to Assess the Effect on Glucose Homeostasis of Two Dose Levels of AZD9567, Compared to Prednisolone, in Adults with Type 2 Diabetes

ClinicalTrials.gov Identifier: NCT04556760

Statistical Analysis Plan: Final 3.0, 28 Oct 2021

# Parexel International AstraZeneca D6470C00005

A Phase 2a Randomised, Double Blind, Multi-centre Study to Assess the Effect on Glucose Homeostasis of Two Dose Levels of AZD9567, Compared to Prednisolone, in Adults with Type 2 Diabetes

**Statistical Analysis Plan** 

**Version: Final 3.0** 

Parexel Project Number: CC

Page 1 of 56

# **SPONSOR SIGNATURE PAGE**

| Approved by: | | |
|--------------|-----------------------------|------|
| | PPD | Date |
| | Global Product Statistician | |
| | AstraZeneca | |

# **TABLE OF CONTENTS**

| 1 | INTRODUCTION | • | 9 |
|---|---|---|---|
| 2 | OBJECTIVES AND ENDPOINTS | | 10 |
| 3 | INVESTIGATIONAL PLAN | | 12 |
| 3.1 | Overall Study Design and Plan. | | |
| 3.2 | Variables associated to the different endpoints. | | |
| 3.2.1 | | | |
| 3.2.2 | | | |
| 3.2.3 | | | |
| 4 | STATISTICAL METHODS | | 21 |
| 4.1 | Data Quality Assurance. | | <b>4</b> 1 |
| 4.2 | General Presentation Considerations | | |
| 4.3 | General Variables | | |
| 4.3.1 | | | |
| 4.3.2 | | | |
| 4.3.2 | | | |
| 4.3.3 | 1 | | |
| 4.4 | Software Programs. | | |
| 4.5 | Study Patients | | |
| 4.5.1 | | | |
| 4.5.2 | | | |
| 4.6 | Analysis Sets | | |
| 4.7 | Demographics and Baseline Characteristics | | |
| 4.8 | Baseline, change from baseline and percentage change from baseline definitions | | |
| 4.9 | Medical History | | |
| | Prior and Concomitant Medications, and other treatments | | |
| 4.11 | | | |
| 4.11. | | | |
| 4.11. | 2 Deaths and Serious Adverse Events | 31 | |
| 4.11. | 3 Clinical Laboratory Evaluation | 31 | |
| 4.11. | | | |
| 4.11. | 5 Morning serum cortisol and ACTH | 32 | |
| 4.12 | Pharmacodynamics and Pharmacokinetics | | |
| 4.12. | | | |
| 4.12. | 1.1 Multi-center Studies | | |
| 4.12. | 1.2 Handling of Dropouts or Missing Data | 33 | |
| | 1.3 Interim Analyses | | |
| 4.12. | | | |
| 4.12. | 3 Pharmacokinetics | 44 | |
| 4.12. | 3.1 Concentrations | 44 | |
| 4.12. | 3.2 Pharmacokinetic Parameters | 45 | |
| 4.13 | Other Analyses | 47 | |
| 4.14 | Determination of Sample Size | 47 | |
| 4.15 | Changes in the Conduct of the Study or Planned Analysis | 48 | |
| 5 | REFERENCES | | 49 |
| 6 | APPENDICES | | 50 |

# Parexel International

| D6470C00005 | | Statistical Analysis Plan |
|---|---|---|
| 6.1 | Schedule of Activities | 50 |
| 6.2 | Blood Sampling Schedule for Mixed Meal Tolerance Tests (MMTTs) | 56 |

# **REVISION HISTORY**

| Version No. | Effective Date | Summary of Change(s) |
|---|---|---|
| D 001 | D 00 2020 | , , |
| Draft 0.1 | Dec 08, 2020 | New document |
| Draft 0.2 | Jan 26, 2021 | Analysis sets redefined, certain sections updated |
| Draft 0.3 | Feb 14, 2021 | Updates based on version 3.0 of the draft Protocol Amendment 2 (dated 10 Feb 2021) |
| Draft 0.4 | March 04, 2021 | Updates based on AZ comments |
| Draft 0.5 | March 12, 2021 | Updates based on AZ comments |
| Final 1.0 | April 28, 2021 | Updated based on PXL and AZ comments |
| Final 1.0 | May 24,2021 | Updated based on PXL and AZ comments during interim analysis n 1. |
| Final 2.0 | Aug 16, 2021 | Removal of figures that are not require for CSR. |
| | | Removed requirement that each cohort should be presented as a separate output. |
| Final 3.0 | Oct 28, 2021 | Update the Statistical Analysis Plan (SAP) to v3.0 in order to re-insert texts which had been included in SAP v1.0 but erroneously had been deleted in SAP v2.0. |
| | | Note: This does not mean a change to the planned analysis but the correction of an error. |

# LIST OF ABBREVIATIONS

| Abbreviation | Explanation |
|---|---|
| ACTH | Adrenocorticotropic hormone |
| AE | Adverse event |
| ALP | Alkaline phosphatase |
| ALT | Alanine transaminase |
| ANOVA | Analysis of variance |
| AST | Aspartate transaminase |
| AUC(0-4) | Area under the curve from zero to 4 hours post-dose |
| AUC(0-6) | Area under the plasma concentration versus time curve from zero to 6 hours post-dose |
| AUC(0-24) | Area under the plasma concentration versus time curve from zero to 24 hours post-dose |
| AUClast | Area under the plasma concentration versus time curve from zero to the last quantifiable concentration |
| CCI | |
| BLQ | Below the lower limit of quantification |
| BP | Blood pressure |
| CfB | Change from baseline |
| CGM | Continuous glucose monitoring |
| CI | Confidence interval |
| CL/F | Apparent total body clearance of drug from plasma after extravascular administration |
| Cmax | Maximum observed drug concentration |
| CRO | Contract Research Organization |
| CRP | C-reactive protein |
| CRU | Clinical Research Unit |
| CSP | Clinical Study Protocol |
| gCSR | Clinical Study Report |
| CSRHLD | Standards for reporting clinical data in a Clinical Study Report or Higher Level Document |
| CV | Coefficient of variation |
| CYP3A4 | Cytochrome P450 3A4 |
| DAS | Disease Activity Score |
| DBP | Diastolic blood pressure |
| DNA | Deoxyribonucleic acid |
| DPP4i | Dipeptidyl peptidase 4 inhibitor |
| ECF | Extracellular fluid |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| EDC | Electronic data capture |

| ENR | All enrolled subjects |
|---|---|
| ET | End of treatment |
| FAS | Full Analysis Set |
| FDA | U.S. Food and Drug Administration |
| FFA | Free fatty acid |
| FGM | Flash glucose monitoring |
| FPG | Fasting plasma glucose |
| FSH | Follicle-stimulating hormone |
| GC | Glucocorticoid |
| GCP | Good Clinical Practice |
| GI | Gastrointestinal |
| GIP | Glucose-dependent insulin releasing polypeptide |
| GLP-1 | Glucagon-like peptide-1 |
| glucose AUC(0-4) | Change in glucose area under the concentration-time curve over 4 hours |
| GMP | Good Manufacturing Practice |
| GR | Glucocorticoid receptor |
| HbA1c | Haemoglobin A1c |
| hCG | Human chorionic gonadotropin |
| HCV | Hepatitis C virus |
| HOMA-IR | Homeostatic model assessment-insulin resistance |
| HOMA-S | Homeostatic model assessment-insulin sensitivity |
| IB | Investigator's Brochure |
| ICH | International Council for Harmonisation |
| ICF | Informed consent form/Intercellular fluid |
| IMP | Investigational medicinal product |
| IPD | Important Protocol Deviation |
| IVRS/IWRS | Interactive Voice/Web Response System |
| LMM | Linear mixed model |
| LPS | Lipopolysaccharide |
| MAD | Multiple ascending dose |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | Mixed model for repeated measures |
| MMTT | Mixed meal tolerance test |
| NC | Not calculable |
| PD | Pharmacodynamic(s) |
| PP | Per Protocol Analysis Set |
| PK | Pharmacokinetic(s) |
| PKAS | PK Analysis Set |

| RA | Rheumatoid arthritis |
|---|---|
| RND | All randomised subjects |
| SAE | Serious adverse event |
| SAF | Safety Analysis Set |
| SAP | Statistical analysis plan |
| SBP | Systolic blood pressure |
| SD | Standard deviation |
| SGLT2i | Sodium-glucose co-transporter-2 inhibitor |
| SGRM | Selective glucocorticoid receptor modulator |
| SoA | Schedule of Activities |
| T2DM | Type 2 diabetes mellitus |
| TBW | Total body water |
| TLFs | Tables, listings and figures |
| TNFα | Tumour necrosis factor alpha |
| t1/2λz | Terminal elimination half-life |
| tmax | Time to reach maximum observed drug concentration |
| ULN | Upper limit of normal |
| U-K | Urinary potassium |
| U-Na | Urinary sodium |
| Vz/F | Apparent volume of distribution following extravascular administration |

#### 1 INTRODUCTION

AZD9567 is a glucocorticoid receptor (GR) modulator that shows promising separation between anti-inflammatory and dysglycaemic effects in preclinical studies and in two dose escalation studies in healthy volunteers (D6470C00001 and D6470C00002). In addition, in a study in patients with active RA (rheumatoid arthritis) (D6470C00003), 40 mg AZD9567 resulted in a similar profile in term of efficacy effects to prednisolone 20 mg following 14 days of once daily dosing. The aim of this study is to assess the effect on glycaemic control of AZD9567 as compared to prednisolone in a more relevant patient population.

The doses used (40 mg AZD9567 [equipotent to 20 mg prednisolone] and 72 mg AZD9567 [equipotent to 40 mg prednisolone]) were chosen based on studies D6470C00001 and D6470C00002 (equipotency was based on ex-vivo lipopolysaccharide [LPS] stimulated tumor necrosis factor alpha [TNFα] release in whole blood). In study D6470C00002, the effect of several doses of AZD9567 up to 80 mg (equipotent to 45 mg prednisolone) on plasma glucose was investigated and compared with prednisolone. After an OGTT (oral glucose tolerance test), the AUC(0-4) (area under the curve) was measured. The result showed that the effect of AZD9567 80 mg on glucose was similar to the lower dose of 5 mg prednisolone despite being equipotent to 45 mg prednisolone.

The analyses described in this SAP (Statistical analysis plan) are based upon the following study documents:

- Clinical Study Protocol Amendment 2 (v3.0), dated 03 March 2021
- Electronic Case Report Form (eCRF), Version 1.0 (October 27, 2020)
- AZ Corporate CSRHLD Reporting Standards v3.3
- The following AZ templates:
  - o AZ Corporate CSRHLD Tables Templates v3.5
  - AZ Corporate CSRHLD Figures Templates v3.2
  - AZ Corporate CSRHLD Listings Templates v1.4
  - o AZ Corporate CSRHLD Reporting Standards v3.3.
  - o AZ Respiratory CSR/HLD Figure Template

This SAP details the statistical methodology to be used for analysing the study data and outlines the statistical programming specifications for the tables, listings and figures (TLFs). It describes the variables and analysis sets, anticipated data transformations and manipulations and other details of the analyses not provided in the Clinical Study Protocol (CSP). The SAP describes the statistical analysis as it is foreseen when the study is being planned if circumstances should arise during the study rendering this analysis inappropriate, or if improved methods of analysis should arise, updates to the analyses may be made in an updated SAP. Any deviations from the SAP after database lock, reasons for such deviations and all alternative or additional statistical analyses that may be performed, will be described in an SAP Addendum and discussed in the Clinical Study Report (CSR).

#### 2 OBJECTIVES AND ENDPOINTS

| Objectives | Endpoints/Outcome measures |
|---|---|
| Primary | |
| To determine the PD effect of AZD9567 on glucose homeostasis compared to prednisolone | Primary endpoint: Change in glucose AUC(0-4) versus baseline compared to prednisolone following a standardised MMTT |
| Secondary | |
| To determine the effect of AZD9567 on CGM compared to prednisolone | <ul> <li>Mean daily glucose at 48 – 72 hours treatment as determined from multiple measures via the CGM system</li> <li>Rise in mean daily glucose over 24-hour periods from start of IMP dosing (0 – 24 hours, 24 – 48 hours, 48 – 72 hours)</li> </ul> |
| To determine the PD effect of AZD9567 following a MMTT compared to prednisolone | <ul> <li>Change from baseline in fasting glucose</li> <li>Change from baseline AUC(0-4) on hormones related to glucose homeostasis (insulin, glucagon, GLP-1, GIP) and FFAs</li> </ul> |

| Objectives | Endpoints/Outcome measures |
|---|---|
| To determine the PD effect of AZD9567 on | Change from baseline in AUC(0-4) |
| glucose homeostasis through an MMTT in | on insulin and C-peptide |
| comparison to prednisolone | |
| To determine the PD effect of AZD9567 on | MMTT derived first phase insulin |
| derived measures of beta cell function from the | response ( $\Delta I_{10}/\Delta G_{10}$ , $\Delta I_{30}/\Delta G_{30}$ , |
| MMTT compared to prednisolone | $\Delta C_{10}/\Delta G_{10}$ , $\Delta C_{30}/\Delta G_{30}$ - where, $\Delta$ : |
| | change from baseline, I: insulin, C: |
| | C-peptide, G: glucose) |
| | Homeostatic model assessment of |
| | insulin resistance (HOMA-IR), |
| | homeostatic model assessment of |
| | insulin sensitivity (HOMA-S) |
| To determine the effect of AZD9567 on U-Na | 24-hour sodium and potassium |
| and U-K excretion compared to prednisolone | concentration |
| To evaluate the PK of AZD9567 following once | Plasma PK parameters |
| daily dosing | Tasma i K parameters |
| To collect plasma samples for analysis of | Plasma concentrations of |
| prednisolone. Reported outside the CSR | prednisolone |
| To explore the relationship between AZD9567 | TNFα concentrations |
| exposure and inhibition of LPS-stimulated TNF $\alpha$ | |
| release for high and low dose comparison | |
| (Cohort 1 and Cohort 2) | |
| Safety | |
| To evaluate the safety and tolerability of | AEs/SAEs |
| AZD9567 compared to prednisolone | Vital signs |
| | • ECGs |
| | Changes in clinical |
| | chemistry/haematology parameters |
| | Morning serum cortisol |
| | • ACTH |

| Objectives | Endpoints/Outcome measures |
|-------------|----------------------------|
| Exploratory | |
| CCI | |
| CCI | |
| CCI | |

#### 3 INVESTIGATIONAL PLAN

### 3.1 Overall Study Design and Plan

This is a randomised, double blind, multi-center, double dummy, two-way cross-over study with the primary objective of determining the effect of AZD9567 on glucose homeostasis (ie, glycaemic control) versus a dose of prednisolone expected to deliver similar anti-inflammatory effects, as assessed by the change in glucose AUC following the standardised mixed meal tolerance test (MMTT) compared to baseline. Approximately 46 participants with type 2 diabetes mellitus (T2DM) will be randomised to achieve 40 evaluable participants completing the study. The study will be conducted in Germany.

AZD9567 will be administered once daily as an oral suspension at two dose levels (40 mg/day and 72 mg/day). Prednisolone capsules will be administered orally at three different dose levels (5 mg/day, 20 mg/day, and 40 mg/day). Since the investigational medicinal product (IMP) has different formulations, it will be administered in a double dummy fashion, with each participant taking both oral suspension and capsules of prednisolone/placebo.

Each cohort will be treated for two 72-hour periods in a cross-over design, with a 3-week Washout period between treatment periods. The total length of participant engagement (from screening D6470C00005 Statistical Analysis Plan

to follow-up) is 79 days; the study duration may be extended for screening and Wash-out (see the Schedule of Activities -SoA-).

There will be three two-way cross-over cohorts, with three different dose combinations (72 mg AZD9567/40 mg prednisolone, 40 mg AZD9567/20 mg prednisolone and placebo/5 mg

1220/30/140 mg predmisolone, 40 mg 1220/30/120 mg predmisolone and placebols mg

prednisolone):

• Cohort 1: participants will be randomised in a ratio of 1:1 to receive AZD9567 and prednisolone

over two 72-hour periods in a cross-over design (72 mg AZD9567 followed by 40 mg

prednisolone [AB sequence group] or 40 mg prednisolone followed by 72 mg AZD9567 [BA

sequence group]). There will be a 3-week Wash-out period between treatment periods. (N = 24)

completed [12 in each sequence group].)

• Cohort 2: participants will be randomised in a ratio of 1:1 to receive AZD9567 and prednisolone

over two 72-hour periods in a cross-over design (40 mg AZD9567 followed by 20 mg

prednisolone [AB sequence group] or 20 mg prednisolone followed by 40 mg AZD9567 [BA

sequence group]). There will be a 3-week Wash-out period between treatment periods. (N = 8

completed [4 in each sequence group].)

• Cohort 3: participants will be randomised in a ratio of 1:1 to receive placebo and prednisolone

over two 72-hour periods in a cross-over design (placebo followed by 5 mg prednisolone [AB

sequence group] or 5 mg prednisolone followed by placebo [BA sequence group]). There will

be a 3-week Wash-out period between treatment periods. (N = 8 completed [4 in each sequence

group].)

With the exception of the SoA, where the headings of visits 4 and 5 include both the day within the

study and within each period (such as 26 and -2 for the same day), all days in this document refer

to days within each period. As an illustration, Day 28 in the study is only referred to as Day 1 in

this document.

In treatment period 1, participants will be fitted with a continuous glucose monitoring/flash glucose

monitoring (CGM/FGM) device on Day -4 on an Out-patient' basis. Within each treatment period,

participants will be admitted to the CRU on Day -2. On Day -1, they will have a baseline MMTT.

Dosing of IMP will occur on Days 1 to 3. The CGM/FGM device will be removed on Day 4.

CCI

Page 13 of 56

Participants will have an MMTT in the morning of Day 4, before being discharged from the CRU in the afternoon of Day 4.

# 3.2 Variables associated to the different endpoints.

As stated in section 3.1, Days refer to those within each treatment period (eg, Days 24, 26, 27, 28, 39, 30, 31 in the study referred to as Day -4, -2, -1, 1, 2, 3 and 4).

# 3.2.1 Pharmacodynamic Variables

## Continuous Glucose Monitoring (CGM)/Flash Glucose Monitoring (FGM)

A CGM/FGM device will be fitted on an Out-patient' basis on Day -4 and removed on Day 4. Mean daily glucose will be determined from multiple measures.

# Mixed Meal Tolerance Test (MMTT)

On Days -1 and 4, a standardised mixed meal (meal should be consumed as fast as the participant can, within 30 minutes) will be administered around 07:00 a.m., after an overnight fast of 12 hours. Blood samples will be taken according to the schedule in section 6.2 for analysis of glucose, insulin, C-peptide, Glucagon-like peptide-1 (GLP-1), Glucose-dependent insulin releasing polypeptide (GIP), glucagon and free fatty acids (FFAs).

### 24-hour Urinary Sodium (U-Na) and Urinary Potassium (U-K)

On Days -1 and 3, sodium and potassium concentrations in urine will be measured over 24 hours.

# TNFα Concentrations

On Day 3, TNF $\alpha$  concentrations in blood will be measured and analysed with and without stimulation with LPS in Cohorts 1 and 2.





# 3.2.2 Safety and Tolerability Variables

# Adverse Events and Serious Adverse Events

Adverse events will be reported by the participant or by a caregiver, surrogate, or the participant's legally authorised representative.

# Time Period and Frequency for Collecting AE and SAE Information

Adverse Events will be collected from time of signature of the informed consent form throughout the treatment period, including the follow-up period, to the Final/ET visit.

Serious adverse events will be recorded from the time of signing of the ICF.

#### Adverse event variables

The following variables will be collected:

- AE (verbatim)
- The date and time when the AE started and stopped
- Maximum intensity of the AE:
  - O Intensity rating scale:

Mild (awareness of sign or symptom, but easily tolerated)

Moderate (discomfort sufficient to cause interference with normal activities)

Severe (incapacitating, with inability to perform normal activities)

- Whether the AE is serious or not
- Investigator causality rating against the Investigational Product(s)
   (yes or no)
- Action taken with regard to Investigational Product(s)
- AE caused participant's withdrawal from study (yes or no)
- Outcome.

In addition, the following variables will be collected for SAEs:

- Date AE met criteria for SAE
- Date investigator became aware of SAE
- AE is serious due to (reason)
- Date of hospitalisation
- Date of discharge
- Probable cause of death
- Date of death
- Autopsy performed
- Causality assessment in relation to Study procedure(s)
- Causality assessment to other medication.

# **Causality Collection**

The investigator should assess causal relationship between Investigational Product and each AE, and answer 'yes' or 'no' to the question 'Do you consider that there is a reasonable possibility that the event may have been caused by the investigational product?'.

For SAEs, causal relationship should also be assessed for other medication and study procedures. Note that for SAEs that could be associated with any study procedure the causal relationship is implied as 'yes'.

## Adverse Events Based on Signs and Symptoms

All AEs spontaneously reported by the participant or reported in response to the open question from the study site staff: 'Have you had any health problems since the previous visit/you were last asked?', or revealed by observation will be collected and recorded in the eCRF. When

Parexel International

D6470C00005 Statistical Analysis Plan

collecting AEs, the recording of diagnoses is preferred (when possible) to recording a list of

signs and symptoms. However, if a diagnosis is known and there are other signs or symptoms

that are not generally part of the diagnosis, the diagnosis and each sign or symptom will be

recorded separately.

Adverse Events Based on Examinations and Tests

Deterioration as compared to baseline in protocol-mandated laboratory values, vital signs

ECGs, and other safety assessments should therefore only be reported as AEs if they fulfil any

of the SAE criteria, are the reason for discontinuation of treatment with the investigational

product or are considered to be clinically relevant as judged by the investigator (which may

include but not limited to consideration as to whether treatment or non-planned visits were

required or other action was taken with the study treatment, eg, dose adjustment or drug

interruption).

If deterioration in a laboratory value/vital sign is associated with clinical signs and symptoms,

the sign or symptom will be reported as an AE and the associated laboratory result/vital sign

will be considered as additional information. Wherever possible the reporting investigator uses

the clinical, rather than the laboratory term (eg, anaemia versus low haemoglobin value). In the

absence of clinical signs or symptoms, clinically relevant deteriorations in non-mandated

parameters should be reported as AE(s).

Any new or aggravated clinically relevant abnormal medical finding at a physical examination

as compared with the baseline assessment will be reported as an AE unless unequivocally

related to the disease under study.

**Physical Examinations** 

A complete examination will include: general appearance, respiratory, cardiovascular,

abdomen, skin, head and neck (including ears, eyes, nose and throat), lymph nodes, thyroid,

muscular-skeletal (including spine and extremities), and neurological systems.

A brief examination will include, at a minimum, assessments of the skin, lungs, cardiovascular

system, and abdomen (liver and spleen).

CCI

## Height and weight

Height and weight will be assessed at the times specified in the SoA. In addition, as detailed in section 3.2.1, weight will be assessed Each time the COI device is used.

## Vital Signs

Vital signs will be assessed after the participant has rested in the supine position for  $\geq 10$  minutes at the times specified in the Schedule of Activities:

- Systolic BP (mmHg)
- Diastolic BP (mmHg)
- Pulse (bpm).

Blood pressure will be measured in triplicate, with all readings averaged to give the measurement to be recorded in the eCRF.

Aural body temperature (°C) will also be measured.

# Electrocardiograms

A 12-lead ECG will be performed after 10 minutes' supine rest at the times specified in the Schedule of Activities. The investigator will interpret the overall results as normal or abnormal and, if abnormal, whether or not it is clinically significant.

The type and nature of abnormalities will be documented whereas clinically significant findings will be recorded as AEs, if applicable.

Additional ECG unscheduled assessments may be performed by the investigator.

As detailed in the eCRF, the following parameters will be assessed in 12-lead ECGs:

RR-interval (msec)

QRS-interval (msec)

QT-interval (msec)

QT-interval corrected using the Fridericia correction formula (QTcF) (msec)

Heart rate (beats per minute [bpm]).

The ECG will be evaluated by the Investigator as 'Normal' or 'Abnormal'.

# Clinical Safety Laboratory Assessments

Blood and urine samples for the determination of clinical chemistry (including triglycerides and HDL-C), haematology, coagulation, urinalysis, and additional laboratory variables (HbA1c [screening only], serum cortisol, ACTH, CCI hCG, 24-hour U-Na and U-K, and FFAs) will be taken.

AEs based on examinations and tests should be reported as described in Section 8.4.5 of the CSP.

# **Laboratory Variables**

| Haematology/Haemostasis (whole blood) | Clinical Chemistry (serum or plasma) |
|---|---|
| White blood cell (WBC) total and differential count | Creatinine |
| Red blood cell (RBC) count | Bilirubin, total and direct |
| Platelet count | Alkaline phosphatase (ALP) |
| Haemoglobin (Hb) | Aspartate transaminase (AST) |
| Haematocrit (HCT) | Alanine transaminase (ALT) |
| Mean corpuscular volume (MCV) | Gamma glutamyl transpeptidase (GGT) |
| Mean corpuscular haemoglobin (MCH) | Potassium |
| Mean corpuscular haemoglobin concentration (MCHC) | Calcium, total |
| Neutrophils (absolute) | Sodium |
| Lymphocytes (absolute) | Uric acid |
| Monocytes (absolute) | Urea |
| Eosinophils (absolute) | Phosphate |
| Basophils (absolute) | Bicarbonate |
| Reticulocytes absolute count | High sensitivity C-reactive protein (hsCRP) |
| Urinalysis | Triglycerides |
| Blood | High-density lipoprotein-cholesterol (HDL-C) |
| Protein | TSH <sup>a</sup> |
| 24-hour sodium and potassium | Serology |
| Glucose | Human immunodeficiency virus (HIV) I and II <sup>a</sup> |
| Creatinine | Hepatitis A virus (HAV) antibody <sup>a</sup> |
| Microscopy (if positive for protein or blood) | Hepatitis B surface antigen (HbsAg) <sup>a</sup> |
| Other | Hepatitis C virus (HCV) antibody <sup>a</sup> |
| COVID-19 polymerase chain reaction (PCR) | Tuberculosis <sup>a</sup> |
| HbA1C <sup>a</sup> | COVID-19 |

#### **Laboratory Variables**

| Glucose (fasting) | Pregnancy testing |
|---|---|
| Insulin | Human-beta chorionic gonadotrophin (hCG) (blood and |
| | urine dipstick) |
| C-peptide | Follicle-stimulating hormone (FSH) (serum) <sup>a, b</sup> |
| Serum cortisol <sup>c</sup> | Coagulation |
| Adrenocorticotropic hormone (ACTH) ° | International normalized ratio (INR) |
| Free fatty acids (FFAs) | Prothrombin time (PT) |
| CCI | Activated partial thrombin time (aPTT) |
| CCI | |

- <sup>a</sup> Screening only.
- b Females only. FSH assessment is for menopausal status.
- Collected from the fasting MMTT blood samples (-15 min) when MMTT is assessed at the same visit. For the MMTT a standardised mixed meal is to be provided around 07:00 on Day -1 and Day 4 (in each period). Serum cortisol, CCI and ACTH are to be collected from the fasting MMTT blood samples, which is -15 minutes prior to the mixed meal on Days -1 and 4 (in each period).

#### 3.2.3 Pharmacokinetic Variables

Pharmacokinetic analysis for AZD9567 will be performed by Covance Clinical Pharmacokinetic Alliance. Pharmacokinetic parameters will be derived using standard non-compartmental methods using WinNonLin version 8.1 or higher (Certara).

The following PK parameters will be calculated:

- AUClast Area under the plasma concentration versus time curve from zero to the last quantifiable concentration
- AUC(0-24) Area under the plasma concentration versus time curve from zero to 24 hours post-dose
- AUC(0-6) Area under the plasma concentration versus time curve from zero to 6 hours post-dose
- Cmax Maximum observed drug concentration

- tmax Time to reach maximum observed drug concentration
- t½λz Terminal elimination half-life
- CL/F Apparent total body clearance of drug from plasma after extravascular administration
- Vz/F Apparent volume of distribution following extravascular administration.

Additional PK parameters may be determined.

The following diagnostic parameters will be listed but not summarised:

- $\lambda z$  lower Lower (earlier) t used for  $\lambda z$  determination
- $\lambda z$  upper Upper (later) t used for  $\lambda z$  determination
- $\lambda zN$  Number of data points used for  $\lambda z$  determination
- $\lambda z$  span ratio Time period over which  $\lambda z$  was determined as ratio of  $t\frac{1}{2}$
- Rsq\_adj Statistical measure of fit for the regression used for  $\lambda z$  determination adjusted for the number of used data points (n obs).

### 4 STATISTICAL METHODS

### 4.1 Data Quality Assurance

TLFs in the report will be checked for consistency, integrity and in accordance with standard Parexel procedures.

#### 4.2 General Presentation Considerations

Summary tables will include the results of each planned sequence in the case of the all randomised subjects set (RND), planned treatment in the case of the Full Analysis Set (FAS) or actual treatment in the case of the Safety Analysis Set (SAF), Per Protocol Analysis Set (PP) and the PK Analysis Set (PKAS).

Non-PK continuous data will be summarised in terms of number of observations, the mean, standard deviation (SD), median, 25th and 75th percentiles (where appropriate), minimum, maximum. In the

Parexel International

D6470C00005 Statistical Analysis Plan

case of PK data, the Pharmacokinetics section of this SAP lists the statistics included in the summary

tables.

For continuous data, the mean, median and geometric mean will be rounded to one additional decimal

place compared to the original data. The SD and geometric coefficient of variation (CV) will be

rounded to two additional decimal places compared to the original data. Minimum and maximum will

be displayed with the same accuracy as the original data. The maximum number of decimal places

reported will be four for any summary statistic.

One decimal will be presented for the geometric CV % included in the PK summary tables.

Categorical data will be summarised in terms of the number of participants, frequency counts and

percentages.

Percentages will be presented to one decimal place. Percentages will not be presented for zero counts.

Percentages will be calculated using n as the denominator (participants included in the analysis sets

or number of non-missing values).

Confidence intervals (CIs) will be presented to one additional place than the original data. P-values

greater than or equal to 0.001, in general, will be presented to three decimal places. P-values less than

0.001 will be presented as "<0.001".

Unless otherwise noted, for the calculation of a change from baseline, the last reliable assessment (in

the case of blood pressure, the average of triplicate assessments) prior to the first dose of each study

treatment will be considered the baseline measurement.

In the case of assessments at scheduled timepoints, the post-baseline scheduled or non-scheduled

reliable assessment closest to the timepoint will be used. If two post-dose assessments are equidistant

from a timepoint, the earlier of the two will be used.

All glucose values will be presented in mmol/L. The following formula will be used for the

conversion of glucose concentrations from mg/dL to mmol/L:

Glucose (mmol/L) = Glucose (mg/dL)  $\times 0.0555$ 

All analyses of pharmacodynamics endpoints involving a linear mixed model will be run separately

for each cohort.

CCI

Change from baseline and percent change from baseline

The change from baseline at each visit will be calculated as:

Change from baseline at visit X = absolute value at visit X-baseline value

The percent change from baseline will be calculated as:

Percent change from baseline = (change from baseline/baseline value) ×100%

If either a visit value or the baseline visit value is missing, the change from baseline value and the percent change from baseline will be set to missing.

#### 4.3 General Variables

# 4.3.1 Study Day Definitions

Study day 1 is defined as the date of first dose of study treatment within each treatment period. Within each treatment period, for visits (or events) prior to first dose, study day is defined as 'date of visit [event] – date of first dose of study treatment'. For visits (or events) that occur on or after first dose of study treatment, study day is defined as 'date of visit [event] – date of first dose of study treatment + 1'.

"Days since last dose" is defined as 'date of visit [event]— date of last dose of study treatment' where "date of last dose" is defined as the date of dosing immediately preceding the event occurrence.

# 4.3.2 Handling of Missing Data

Unless otherwise stated, missing data will not be imputed.

4.3.2.1 Imputations of Partial Medication and AEs Dates

There will be no imputation of any incomplete dates.

The following rules will be used to determine whether or not an AE has taken place on-treatment:

- 1. An AE starting from last dose plus 21 days will be considered on-treatment.
- 2. An AE with an incomplete start date and whose end date is not prior to the time of dosing on Day 1 will be considered to have taken place on-treatment unless the non-missing components of the incomplete start date indicate that the start date falls outside the time from dosing on Day 1 to last dose plus 21 days.

D6470C00005 Statistical Analysis Plan

The following rules will be used to assign concomitance to a medication:

1. Exclusively prior medications are those that started and stopped prior to the first dose of the

investigational medicinal product (IMP) in the first treatment period and those that started

and stopped after 21 days after the last dose in the first period and before the first dose of

IMP in the second period. Medications taken between the first dose and up to 21 days after

the last dose in any period are concomitant (including medications that started prior to dosing

and continued after)

2. A medication with incomplete start and/or end dates will be considered concomitant unless

the non-missing components of the incomplete dates indicate that the intake of the medication

did not take place between Day 1 and the last dose plus 21 days.

AEs and medications with completely missing end dates will be assumed to be ongoing.

4.3.3 Imputation Rules for Laboratory Values Outside of Quantification Range

Values of the form "< x" (i.e., below the lower limit of quantification [LLoQ]) or "> x" (i.e., above

the upper limit of quantification [ULoQ]) will be imputed as "x" in the calculation of summary

statistics but displayed as "< x" or "> x" in the listings.

4.4 Software Programs

All report outputs will be produced using SAS® version 9.4 in a secure and validated environment.

PK analyses will be produced using Phoenix® WinNonLin (WNL) version 8.1 or later in a secure

and validated environment.

All report outputs will be provided to the Sponsor. Tables and figures will be combined in one PDF

document and listings in another.

4.5 Study Patients

4.5.1 Disposition of Patients

A listing will be created for subjects discontinued from the study using the ENR. An additional

listing will be created for subjects completing the study using the RND. Both listings will include

the standardised disposition term and the date of disposition event.

CCI

D6470C00005 Statistical Analysis Plan

A summary table will be created and will include, in addition to the number of patients enrolled, the number and percentage of patients who:

- were randomised
- were not randomised
- received at least a dose of the first treatment
- completed the first treatment
- discontinued the first treatment
- received at least a dose of the second treatment
- completed the second treatment
- discontinued the second treatment
- completed study
- were withdrawn from the study for any reason (one row in the table for all reasons)
- were withdrawn from the study for <u>each</u> reason (one row in the table for each reason).

#### 4.5.2 Protocol Deviations

Important protocol deviations (IPD) may lead to the exclusion of participants from the PP and the PKAS. Deviations will be defined before database lock. Important deviations will include the following:

- Violation of inclusion and/or exclusion criteria
- Administration of prohibited concomitant medications expected to influence the primary endpoint
- Receiving incorrect study intervention than randomised to.

All protocol deviations will be discussed at a data review meeting prior to database lock in order to define the analysis sets for the study. All IPDs will be listed by participant.

The Protocol Deviation Specifications will be followed to assess which protocol deviations are important in a Data Review Meeting (DRM) shortly before database lock/unblinding. A DRM report detailing the assessment of protocol deviations, AEs, the assignment of participants to analysis sets and the exclusion of data from specific analyses will be signed by all scientific experts.

The number and percentage of patients in the FAS meeting each IPD criterion will be summarised by cohort. Patients deviating from an IPD more than once will be counted once for that criterion. Any patients who have more than one IPD will be counted once in the overall summary.

The number of enrolled patients included/excluded from each of the analysis sets will be summarised. Patients and data excluded from each analysis set will be listed with the reason (such as the specific IPDs or AEs) for exclusion.

# 4.6 Analysis Sets

The following sets are defined:

| Population/Analysis set | Description |
|---|---|
| All enrolled subjects (ENR) | All participants who signed informed consent prior to any study-related procedures. |
| All randomised subjects (RND) | All participants in the ENR randomised to one of the two sequence groups within a cohort. The ENR will be analysed according to the planned sequence or treatment. |
| Full Analysis Set (FAS) | All participants in the RND who received at least one dose of study intervention. The FAS will be analysed according to the planned treatment and will be used as the primary population for reporting pharmacodynamic data and to summarize baseline characteristics. Any important deviations from randomised treatment will be listed and considered when interpreting the pharmacodynamic data. |
| Safety Analysis Set (SAF) | All participants in the RND who received at least one dose of study intervention. The SAF will be analysed according to the actual treatment. |
| Per Protocol Analysis Set (PP) | All participants in the FAS who did not have an important protocol deviation considered to have an impact on the analysis of the primary endpoint and who completed the study. The PP will be analysed according to the actual treatment received. |
| PK Analysis Set (PKAS) | All participants in the FAS with at least one quantifiable AZD9567 concentration and no important protocol deviations, or AEs considered to have an effect upon PK. Participants may be excluded from the PK population if they have an AE of vomiting before 2x the median tmax of the group. The PKAS will be analysed according to the actual treatment. |

# 4.7 Demographics and Baseline Characteristics

Demographic characteristics (age, sex, race, ethnicity, country) and baseline patient characteristics (height, weight and BMI) will be listed and will be summarised by cohort in the SAF and FAS. In

Parexel International

D6470C00005 Statistical Analysis Plan

addition to presenting descriptive statistics for age, the summary table will present the number and

percentage of patients per age group (18-44, 45-64 and 65-75 years).

4.8 Baseline, change from baseline and percentage change from baseline definitions

Demography and baseline characteristics

For demography and baseline characteristics other than weight, the baseline will be the assessment

at screening. For weight, the baseline will be the assessment at Day -1 performed by means of the

device. If the weight at Day -1 is missing, the weight at Day -2 (or at Screening, in the case of

period 1 if the value at Day -2 is also missing) will be the baseline for such a period.

**Pharmacodynamics** 

Change in AUC(0-4)

In the case of the linear mixed models for the change from baseline in glucose AUC(0-4) (primary

endpoint), hormones related to glucose homeostasis (insulin, glucagon, GLP-1, GIP), FFAs and C-

peptide (secondary endpoints), the baseline measurement will be the AUC(0-4) on Day -1 (i.e., prior

to first dosing) of each period.

Glucose concentrations assessed by CGM

For the calculation of the rise in mean glucose and the mean daily glucose, the baseline will be the

average of the values from -24 hours to first dosing on Day 1 (values from -72 to -24 hours will be

excluded from the baseline) of each period.

For the MMRM for the rise in mean glucose and the mean glucose, the baseline included as a

covariate in the model will be the value -24 hours to first dosing on Day 1 of each period.

MMTT derived first phase insulin response

For the calculation of the change from baseline of insulin, glucose and C-peptide included in the

calculation of  $\Delta I10/\Delta G10$ ,  $\Delta I30/\Delta G30$ ,  $\Delta C10/\Delta G10$  and  $\Delta C30/\Delta G30$ , the baseline will be value at

Day -1 of each period.

D6470C00005 Statistical Analysis Plan

### 24-hour U-Na and U-K

For Na and K and the Na/K ratio, the baseline will be the value at Day -1 in each period.



# <u>Safety</u>

# ECG and vital signs

For ECG and vital signs, the baseline will be the pre-dose assessment at Day 1 in each period. If this value is missing the value closest in time prior to Day 1 within the same visit (or at Screening, in the case of period 1) will be the baseline for such a period.

# Clinical chemistry/haematology/urinalysis

For the safety laboratory assessments, the baseline for the calculation of the change from baseline will be the pre-dose assessment at Day 1 in each period. If this value is missing, the value closest in time prior to Day 1 within the same visit (or at Screening, in the case of period 1) will be the baseline for such a period.

For the linear mixed models for Na, K and Na/K, the baseline included as covariate will be the same as that used to calculate the change from baseline.



D6470C00005 Statistical Analysis Plan

CCI

### Serum cortisol and ACTH

For the calculation of the difference in the concentration of each of these hormones between Days -1 and 4 of each period, the baseline will be value on Day -1. If the concentration of ACTH at Day -1 in period 1 is missing, the concentration at the Screening visit will be the baseline for such a period.

# 4.9 Medical History

The Full Analysis Set will be used for the presentation of the data.

Medical history data will be listed by patient.

A summary of the number and percentage of patients with any relevant medical history will be presented by SOC and PT, by treatment sequence.

Relevant surgical history will be listed in the same manner.

Medical history data of diabetes will be listed by patient including start date and end date or on going.

#### 4.10 Prior and Concomitant Medications, and other treatments

All listings and tables will be based on the Safety Analysis Set.

Medications will be coded using the World Health Organisation-Drug Dictionary (WHODRUG) and will be classified by Anatomical Therapeutic Chemical (ATC) categories.

Exclusively prior medications are those that started and stopped prior to the first dose of the investigational medicinal product (IMP) in the first treatment period and those that started and stopped after 21 days after the last dose in the first period and before the first dose of IMP in the second period. Medications taken between the first dose and up to 21 days after the last dose in any period are concomitant (including medications that started prior to dosing and continued after).

Concomitant medication will be listed by participant and will include the reported name, anatomical therapeutic chemical (ATC), route of administration, total dose, frequency, start date/time, duration, whether or not ongoing and indication and will be summarised by ATC and PT.

Parexel International

D6470C00005 Statistical Analysis Plan

Medications ongoing during both the periods will be counted under both Period 1 and Period 2.

Prior and concomitant use of Metformin will be listed by participant and will include the total dose,

frequency, start date/time, duration and whether or not ongoing and will be summarised by ATC

and PT.

The number of subjects taking concomitant medications under each treatment will be summarised

by ATC classification/ Generic term.

The duration will be calculated as:

Duration (in days) = (end date - start date) + 1, if only date is known.

4.11 Safety and Tolerability Evaluation

The actual treatment will be used for all safety and tolerability analyses. All listings and tables will

be based on the Safety Analysis Set.

The listings of the safety data (AEs, laboratory data, vital signs, and ECG) will include scheduled

and unscheduled assessments.

4.11.1 Adverse Events

Within each cohort, AEs will be assigned as having taken place after each of the two treatments if

the start of the AE is after the first dose of the treatment but before the end of 21 days after the last

dose (i.e., the end of Day 24, in the case of subjects whose last dose was on Day 3). AEs on Day 1

with a missing start time will be assumed to have started after the first dose.

In order to assign the corresponding SOC and preferred term to each AE, AEs will be coded using

the Medical Dictionary for Regulatory Activities (MedDRA) Version 22.1 or higher.

AEs occurring prior to the time of dosing on Day 1 and after 21 days after the last dose will not be

included in summaries.

An AE listing for the Safety analysis set will cover details for each individual AE. A summary table

with the number of AEs, by SOC and PT will be created.

The following summaries for the number and percentage of participants will be created:

CCI

- Number of subjects with adverse events in any of these categories:
  - Any AE
  - Any AE with outcome = death
  - Any SAE (including events with outcome = death)
  - Any AE leading to discontinuation of IP
  - Any AE leading to drug interruption
  - Any AE leading to withdrawal from study
- Number of subjects with adverse events, by SOC and PT
- Number of subjects with adverse events, by PT
- Number of subjects with adverse events leading to discontinuation of investigational product, by system organ class and preferred term.

In summaries including SOC or PT, the summaries will first be sorted by decreasing percentage of participants in each SOC and PT within SOC, and then alphabetically by SOC, and PT within SOC.

The following summaries for the number and percentage of adverse will be created:

• Number of adverse events by system organ class and preferred term.

#### 4.11.2 Deaths and Serious Adverse Events

The number of SAEs, by SOC and PT will be summarised.

These summaries will be created for the number of subjects and adverse events, by SOC and PT.

# 4.11.3 Clinical Laboratory Evaluation

All values will be classified as low (below range), normal (within range), or high (above range) based on central laboratory reference ranges.

The Na/K ratio will be calculated at each timepoint and this ratio will be included in clinical chemistry listings and tables. All clinical laboratory results will be listed.

The comparison of the effect of treatment on changes in Na, K and Na/K will be analysed by means of the same statistical model as that used for the analysis of the primary endpoint.

For haematology, clinical chemistry and coagulation a table with descriptive statistics of absolute values and changes from baseline for each laboratory variable over time. Only planned tests will be summarized. In the case of the urinalysis, individual measurements will be listed and a summary table

D6470C00005 Statistical Analysis Plan

of the baseline versus maximum value on-treatment (ie, a shift table) will be created.

The on-treatment definition will be based on the on-treatment definition used for AE.

4.11.4 Vital Signs, ECGs

Vital Signs

Vital signs data will be listed by participant including changes from baseline. Flags for a clinically

significant assessment will be provided in the listing.

Descriptive statistics for absolute values and changes from baseline will be presented by treatment

and by cohort.

**ECGs** 

All ECG parameters will be listed by participant including changes from baseline for numeric ECG

parameters. Abnormalities in ECG will also be listed.

Descriptive statistics for absolute values and changes from baseline will be presented by treatment

and cohort. The on-treatment definition will be based on the on-treatment definition used for AE.

The number and percentage of participants under each treatment exceeding the following ICH

boundaries of QTcF will be tabulated:

• Absolute value > 450 msec and > 480 msec

• Increase from baseline > 30 msec and > 60 msec.

This summary table will also include the number and percentage of participants under each treatment

exceeding the following values:

• Absolute value >450 msec and Increase from baseline >30 msec

• Absolute value >500 msec and Increase from baseline >60 msec.

The following figure will be provided for each ECG parameter:

- Box-plot by treatment and day

4.11.5 Morning serum cortisol and ACTH

The morning serum cortisol and ACTH will be listed and tables with descriptive statistics for the

value -15 minutes prior to the mixed meal on Days -1 and 4 (in each period) and change from baseline

will be created.

CCI

# 4.12 Pharmacodynamics and Pharmacokinetics

### 4.12.1 Analysis and Data Conventions

This study aims to demonstrate that AZD9567 improves glucose homeostasis compared to oral prednisolone.

The null hypothesis for the primary analysis is:

H<sub>0</sub>: there is no difference in the change in glucose AUC(0-4) versus baseline in AZD9567 compared to prednisolone following a standardised MMTT.

The alternative hypothesis for the primary analysis is:

H<sub>a</sub>: there is a difference in the change in glucose AUC(0-4) versus baseline in AZD9567 compared to prednisolone following a standardised MMTT.

In order to test the null hypothesis, a main analysis involving the FAS will be conducted. If more than 10% of participants receive the wrong treatment, a sensitivity analysis involving the PP will be conducted.

The following comparison will be performed:

- 72 mg AZD9567 versus 40 mg prednisolone (Cohort 1)
- 40 mg AZD9567 versus 20 mg prednisolone (Cohort 2)
- Placebo versus 5 mg prednisolone (Cohort 3)

As this is a Phase 2a study, no adjustments for multiple testing will be performed.

#### 4.12.1.1 Multi-center Studies

No adjustments for center will be performed.

### 4.12.1.2 Handling of Dropouts or Missing Data

Summary statistics will be based on non-missing values.

#### 4.12.1.3 Interim Analyses

Two interim analyses are planned.

Parexel International

D6470C00005 Statistical Analysis Plan

The first interim analysis will be conducted when 50% of the participants in Cohort 1 have completed

the study. The purpose of the first interim analysis is to evaluate the feasibility of the assumptions

and conduct sample size re-estimation if required.

The main objective of the first interim analysis is to report the statistical analyses involving the first

endpoint, the secondary endpoints related to glucose (mean daily glucose at 48-72 hours treatment

and rise in mean daily glucose over 24-hour periods from start of IMP dosing) and the safety

endpoints (AEs/SAEs) for 50% of the subjects in Cohort 1.

The second interim analysis will be conducted when all the participants in Cohort 1 have completed

the study. The main objective of the second interim analysis is to report the statistical analyses

involving all subjects in Cohort 1.

The second interim analyses will not include PK data.

4.12.2 Pharmacodynamics

All the models presented in this section will be analysed with unstructured covariance structure used

for the within-participant errors. In the case of a model which does not converge, the analysis will be

performed with a Toeplitz covariance structure and, in case of non-convergence, it will be performed

with a compound symmetry structure.

Primary endpoint

The primary endpoint is the change in glucose AUC(0-4) and will be summarised by timepoint

(baseline and Day 4) and by each cohort. The comparison of the change in glucose AUC(0-4) (where

change from baseline in glucose AUC is assumed to be normally distributed) between the two

treatments administered within each cohort after a standardised MMTT will be performed by means

of two linear mixed effects models, with an unstructured covariance structure, with treatment, period

and sequence as fixed effects, participant within sequence as random effect and baseline as covariate.

Two models will be run separately for each cohort:

1. In the first model, the dependent variable will be the change from baseline in AUC(0-4)

whereas the AUC(0-4) on Day -1 will be included as a covariate. The treatment effects will

be estimated by the Least Square means (LS means) and their 95% CIs and the difference

between the two treatments by the difference in LS means with its 95% CI.

CCI

- 2. The second model will involve the following three steps:
  - a) Log-transformation of the AUC(0-4):

First, the AUC(0-4) in Day -1 and the AUC(0-4) in Day 4 will be log-transformed. The log-transformed AUC(0-4) in Day -1 will then be subtracted from the log-transformed AUC(0-4) in Day 4 to calculate the change in AUC (0-4) in log units.

- b) Execution of the model:
  - The model will include the change in AUC (0-4) in log units as a dependent variable and the log-transformed AUC(0-4) in Day -1 as covariate.
- c) Back-transformation of the results from the model:

The results from the execution of the model will be back transformed to the original scale after an exponentiation of the means and CIs estimated by the model to obtain the percentage geometric LS means of the treatments and their percentage SEs. The LS mean difference and its CI between the two treatments will also be back-transformed to yield the percentage geometric mean ratio between the two treatments with its 95% CI at Day 4.

The statistics for the percentages geometric LS means, percentage SE, percentage geometric LS mean ratio and percentage 95% CI will be calculated as follows:

- i) Percentage geometric LS mean = (exp(estimate)-1)\*100 where estimate is the natural log of LS mean
- ii) Percentage  $SE = sqrt(exp(2*estimate)*SE^2)*100$
- iii) Percentage geometric LS mean ratio= (exp(estimate)-1)\*100 where estimate= log LS mean difference
- iv) percentage 95% CI lower and upper: (exp(lower)-1)\*100; (exp(upper)-1)\*100.

If more than 10% of participants are treated erroneously, a sensitivity analysis will be carried out using the actual treatment received instead. Descriptive statistics and graphical presentations will be presented.

The following graphs will be provided:

- Line plot: the Mean glucose levels (MMTT) by sampling time in minutes by treatment -visit day; (per cohort)
- AUC(0-4) change from baseline (MMTT) for glucose level by visit day of linear mixed model (Full Analysis Set) (all cohorts in a single plot)
- AUC(0-4) percentage change from baseline (MMTT) for glucose level by visit day linear

mixed model (Full Analysis Set) (all cohorts in a single plot).

The following comparison will be performed by the execution of a linear mixed effects model in

each case:

- 72 mg AZD9567 versus 40 mg prednisolone (Cohort 1)

- 40 mg AZD9567 versus 20 mg prednisolone (Cohort 2)

- placebo versus 5 mg prednisolone (Cohort 3).

Secondary endpoints

Mean daily glucose at 48-72 hours (CGM)

The Mean daily glucose (CGM) as well as the change from baseline will be summarize by timepoint

(baseline, 00-24 h, 24-48 h and 48-72 h) and by treatment group.

The comparison of the effect of the two treatments on the mean daily glucose at 48-72 measured by

CGM will be analysed by means of repeated measures mixed model (MMRM) with treatment + time

(0-24h, 24-48h, 48-72h), treatment\*time, period and sequence as fixed effects with baseline (mean

glucose at -24-0 hours) as covariate and participants within sequence as random effect. Two models

will be run separately for each cohort and will be:

1. In the first model, the dependent variable will be the mean daily glucose whereas the mean

glucose at -24-0 hours will be included as covariates. The treatment effects will be estimated

as described in the first model for the primary endpoint.

2. The second model will involve a log-transformation of both the mean glucose at 0-24, 24-

48 and 48-72 hours and the mean glucose at -24-0 hours will be included as a covariate. The

treatment effects will be estimated as described in the second model for the primary endpoint.

The following graphs will be provided:

- Glucose mean levels (CGM) at 0-72 h by treatment (per cohort)

- Glucose mean levels (CGM) at 0-72 h by treatment (all cohorts in a single plot).

Rise in mean glucose at 00-24 h, 24-48h and 48-72 h (CGM)

The comparison of the effect of the two treatments on the rise in mean glucose at 0-24, 24-48 and

48-72 hours will be performed following two different approaches:

CCI

- 1) In the first approach three different models will be performed:
- i) Change at 00-24 h from baseline (24 hours of CGM prior to dosing) performed by means of mixed models with treatment, period and sequence as fixed effects, participants within sequence as random effect and baseline mean glucose
- ii) Change at 24-48 h from baseline (24 hours of CGM prior to dosing) performed by means of mixed models with treatment, period and sequence as fixed effects, participants within sequence as random effect and baseline mean glucose
- iii) Change at 48-72 h from baseline (24 hours of CGM prior to dosing) performed by means of mixed models with treatment, period and sequence as fixed effects, participants within sequence as random effect and baseline mean glucose.
- 2) In the second approach three different models will be performed:
- i) Change at 00-24 h from baseline (24 hours of CGM prior to dosing) performed by means of mixed models with treatment, period and sequence as fixed effects, participants within sequence as random effect and baseline mean glucose
- ii) Change at 24-48 h from baseline (00-24 h) performed by means of mixed models with treatment, period and sequence as fixed effects, participants within sequence as random effect and baseline mean glucose
- iii) Change at 48-72 h from baseline (24-48h) performed by means of mixed models with treatment, period and sequence as fixed effects, participants within sequence as random effect and baseline mean glucose.

The three models for each of the approaches were repeated considering the log-transformation of the dependent variable to obtain the Geometric LS means and the Geometric LSMean Ratio (%).

The following comparison will be performed for the change and the percent change from baseline at 0-24, 24-48 and 48-72 hours:

- 72 mg AZD9567 versus 40 mg prednisolone (Cohort 1)
- 40 mg AZD9567 versus 20 mg prednisolone (Cohort 2)
- placebo versus 5 mg prednisolone (Cohort 3).

The following graphs will be provided:

- Rise in mean change from baseline (CGM) for glucose by Days (Day -1 (24 h prior to dosing), Day 1 (00-24 h), Day 2(24-48 h), Day 3(48-72 h)) 1<sup>st</sup> approach (per cohort)

- Rise in mean change from baseline (CGM) for glucose by Days (Day -1 (24 h prior to dosing), Day 1 (00-24 h), Day 2(24-48 h), Day 3(48-72 h)) 2<sup>nd</sup> approach (all cohorts in a single plot)
- Rise in mean percentage change from baseline (CGM) for glucose by Days (Day -1 (24 h prior to dosing), Day 1 (00-24 h), Day 2(24-48 h), Day 3(48-72 h)) 2<sup>nd</sup> approach (all cohorts in a single plot).

# Change from baseline in fasting glucose

The comparison of the effect of the two treatments on the change from baseline in fasting glucose (-15 minutes) between Days -1 and 4 will be performed by the same model as that for the comparison of the primary endpoint.

The following comparison will be performed for the change and the percent change from baseline at Day 4:

- 72 mg AZD9567 versus 40 mg prednisolone (Cohort 1)
- 40 mg AZD9567 versus 20 mg prednisolone (Cohort 2) placebo versus 5 mg prednisolone (Cohort 3).

### Changes in in AUC(0-4) in hormones, FFAs and C-peptide in response to a MMTT

The comparison of the effect of treatment on changes in insulin, glucagon, GLP-1, GIP, FFAs and C-peptide will be analysed as the primary endpoint.

The following graphs will be provided for each of the variable with the exception of C-peptide:

- The changes from baseline at different timepoints by treatment (all cohorts in a single plot)
- The percentage changes from baseline at different timepoints by treatment (all cohorts in a single plot).

### MMTT derived first phase insulin response

The ratio between variables will be calculated based on the following steps:

i) Calculate  $\Delta$ I10= difference in I (insulin) values between 10 and 0 minutes at Day -1 and Day 4 of each period

- ii) Calculate  $\Delta G10$ = difference in G (glucose) values between 10 and 0 minutes at Day-1 and Day 4 of each period
- iii) Calculate the ratio  $\Delta I10/\Delta G10$  at Day-1 and Day 4 of each period.

The same steps i) to iii) accordingly to timepoints 10 and 30, will be performed for  $\Delta C10/\Delta G10$ ,  $\Delta I30/\Delta G30$ , and  $\Delta C30/\Delta G30$ .

The comparison of the effect of the two treatments on the change in  $\Delta I10/\Delta G10$  and  $\Delta I30/\Delta G30$ , between Days -1 and 4 will be performed by the same model as that for the comparison of the primary endpoint.

The following comparison will be performed for the change from baseline and the percent change from changes from baseline at Day 4 at 10 and 30 minutes:

- 72 mg AZD9567 versus 40 mg prednisolone (Cohort 1)
- 40 mg AZD9567 versus 20 mg prednisolone (Cohort 2)
- placebo versus 5 mg prednisolone (Cohort 3).

The previous analyses will be repeated for the comparison of the effect of the two treatments on the change in  $\Delta C10/\Delta G10$ ,  $\Delta C30/\Delta G30$  using C-peptide instead of insulin in the calculation of these ratios.

### **HOMA-IR and HOMA-S**

A summary of the baseline HOMA-IR and HOMA-S and at Day 4 as well as change from baseline, will be provided by treatment.

### 24-hour U-Na and U-K

The 24-hour Na and K concentration and its ratio (Na/K) in urine will be analysed as the primary endpoint.

The following comparisons will be performed for the change and percentage change from baseline at 0-24 hours on Day 3:

- 72 mg AZD9567 versus 40 mg prednisolone (Cohort 1)
- 40 mg AZD9567 versus 20 mg prednisolone (Cohort 2)
- placebo versus 5 mg prednisolone (Cohort 3).

## TNFα concentrations

Descriptive statistics will be tabulated for the individual measurement points of the LPS-stimulated  $TNF\alpha$  levels.

An ANOVA model with treatment, sequence and subject as random effect will be run separately for each cohort (Cohort 1 and Cohort 2) for the comparisons of the treatments at Day 3.

A scatter plot of individual plasma concentrations of AZD9567 (nmol/L) in a log scale on the X axis versus individual LPS-Stimulated TNFα Levels (ng/L) in log scale on the Y axis will be created.

| CCI | |
|-----|---|
| | _ |



### Calculations of endpoints analysed by statistical models

Calculation of changes from baseline AUC (0-4)

The calculation of the change in glucose, insulin, C-peptide GLP-1, GIP, glucagon and FFAs AUC(0-4) will involve the following steps:

1. The AUC(0-4) each day when the MMTT is consumed will be calculated by means of the linear-log trapezoidal method, i.e., using the linear trapezoidal method when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing.

Accordingly, for a given time interval  $(t_1 - t_2)$ , the AUC could be calculated as follows:

i) by the linear trapezoidal method:

$$AUC = 1/2 (C_1 + C_2) (t_2 - t_1)$$

ii) by the logarithmic trapezoidal method:

AUC = 
$$[(C_1 - C_2)/(\ln(C_1) - \ln(C_2))](t_2 - t_1)$$

where:

C<sub>1</sub> and C<sub>2</sub> are the concentrations at times 1 (t<sub>1</sub>) and 2 (t<sub>2</sub>).the first time interval (t<sub>1</sub> - t<sub>2</sub>) is equal to t<sub>1</sub> (ie, the concentration at -15 minutes is assumed to be the same as if it had been made at 0 minutes),

- for assessments at 10, 20, 30, 60, 75, 120 and 180 minutes, t<sub>1</sub> and t<sub>2</sub> are actual times,
- for the planned assessment at 240 minutes, the planned time (240) will be used if such an assessment has been performed within the allowed time window (±5 minutes).

The total AUC between 0 and 240 minutes will be calculated as the sum of the AUC for each of the intervals described in i) and ii).

The total AUC between two time points will be calculated as the sum of the AUCs calculated for each of the intervals between the two time points.

2. The change in AUC(0-4) will be calculated as:

$$\triangle$$
 AUC(0-4) =AUC(0-4) at Day 4 - AUC(0-4) at Day -1

For the calculation of MMTT  $AUC_{0.4hr}$ , the pre-meal measurement (at -15 min) value will be treated as the value at the meal time (0 minutes). The actual time span for each post-meal measure will be calculated starting from the meal time (0 minutes). If any actual sample collection times are missing, use the scheduled nominal times with reference to the actual meal time to impute.

If the actual sampling times differ from the nominal times more or equal to | 5| min, this will be deemed on case-by-case basis if should be considered protocol deviation.

If greater than 50% of scheduled measures are missing, the AUC will be set as missing; if the first two or last two scheduled measures are both missing, then the AUC will also be set as missing; otherwise:

## For all the MMTT endpoints (glucose, insulin, glucagon, GLP-1, GIP, FFAs and C-peptide):

If any interior measures are missing, the trapezoid rule can be used to calculate the AUC by ignoring the missing time point: i.e. The missing timepoint X will be imputed with the value obtained considering the linear interpolation between the last actual assessment taken prior to point X, and the first actual assessment taken after point X.

For glucose MMTT endpoint:

- If the pre-meal value is missing, set the missing value = 92% of the value for next scheduled time point.
- If the last value is missing, set the missing value = 87% of the value for the time point that is scheduled immediately prior to the last time point.

# For the rest of MMTT endpoints (insulin, glucagon, GLP-1, GIP, FFAs and C-peptide):

- If the pre-meal value is missing, set AUC = missing
- If the last value is missing, set AUC = missing

AUC(0 -4h) calculation assumes that measurements are available at 240 min exactly. Deviation from 240 min will induce a systematic overestimation of the actual value of the sampling time is used exceeds 240 min and underestimation of the actual time is under 240 min. If the deviation is within the allowance window ( $\pm$  5 min) the sampling time will be equated to 240 min. If the sampling time for the 240 min measurement is out of the sampling window ( $\pm$  5 min) a linear interpolation will be considered to assess the value at 240 min using the actual sampling times for the 180 min and the 240 min measurements.

Actual time point (at 180 min) and the time point for last sampling will be defined with  $t_{180}$  and with  $t_{last}$  respectively, and the values of the endpoint (glucose, insulin etc) at the actual measured timepoint and at time point for the last sampling will be defined with  $y_{180}$  and  $y_{last}$ . From the available information ( $t_{180}$ ,  $y_{180}$ ), ( $t_{last}$ ,  $y_{last}$ ) the value at  $t_{240}$ , i.e. the value that the endpoint would have if we would have taken the sample at exactly 240 min form start will be interpolated. Interpolation assumes a linear equation with slope

$$m = (y_{last}-y_{180})/(t_{last}-t_{180})$$

and intercept

$$b = mean(y_{last}; y_{180}) - m*mean(t_{last}; t_{180})$$

giving the value at 240 minutes of:

$$y240 = b + m*240$$
.

The 92 % and 87 % correction factors were based on the MEDI0382 (D5670C00007) study.

## Calculation of HOMA-IR

The HOMA-IR will be calculated as follows based on glucose and insulin measured prior to MMTT (-15 min):

$$HOMA - IR = \frac{Glucose\left(\frac{mmol}{L}\right) \times Insulin\left(mU/L\right)}{22.5}$$

HOMA-S will be calculated as the reciprocal of HOMA-IR.

### 4.12.3 Pharmacokinetics

#### 4.12.3.1 Concentrations

Plasma concentrations of AZD9567 will be listed by actual and relative (to dose administration) sampling time. The following summary statistics will be presented for these concentrations at each time point by treatment and cohort:

- n below the lower limit of quantification (LLOQ) (only for concentrations)
- Geometric Mean
- Geometric CV%
- Geometric Mean SD
- Geometric Mean + SD
- Arithmetic Mean
- Arithmetic SD
- Median
- Minimum
- Maximum

In listings, concentrations less than the lower limit of quantification (LLOQ) will be presented as below the lower limit of quantification (BLQ). In listings and tables where the terms BLQ or LLOQ are included, the LLOQ (numerical value) will be included in a footnote.

For the calculation of statistics, concentrations that are BLQ will be handled as follows at each time point:

- If ≤50% of the concentrations are BLQ, all BLQ values will be set to the LLOQ, and all descriptive statistics will be calculated.
- If >50%, but not all, of the concentrations are BLQ, the arithmetic mean, arithmetic CV, arithmetic mean, and arithmetic SD will be reported as 'NC' (not calculable). The maximum value will be reported from the individual data, and the minimum and median will be set as 'BLQ'.
- If all concentrations are BLQ, no descriptive statistics will be calculated. 'NA' (not applicable) will be presented for geometric CV, and arithmetic SD, and 'BLQ' will be presented for geometric mean, arithmetic mean, median, minimum, and maximum.

Parexel International

D6470C00005 Statistical Analysis Plan

For PK concentration and parameter data, if there are <3 values available at a time point, only the

maximum, minimum, and n will be reported; the remaining descriptive statistics will be reported as

'NC'. Concentrations that are BLQ are considered a value.

Post-dose concentrations where the actual time deviation deviates more than 10% from the scheduled

time will be excluded from summaries by planned time point.

Missing samples will be reported as no sample ("NS") and excluded from analysis.

Source data shall be used in all derived PK concentrations without prior rounding

The following figures, will be generated for each IMP by Cohort:

• Individual Subject Profiles, Plasma Concentration-time Data - Linear Scale: both days on 1

plot

Individual Subject Profiles, Plasma Concentration-time Data - Semi-Logarithmic Scale:

both days on 1 plot

• GMean, Plasma Concentration-time Data - Linear Scale: both days on 1 plot

• GMean, Plasma Concentration-time Data - Semi-Logarithmic Scale: both days on 1 plot.

In combined figures displaying subject profiles, all subjects will be included in the same figure and

concentrations will be displayed by actual sampling time. In figures displaying mean concentrations,

mean concentrations will be displayed by time point.

4.12.3.2 Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated following these guidelines:

Pharmacokinetic analysis will, where possible, be calculated using times recorded in the raw data. If

actual times are missing, nominal times may be used.

The concentrations reported by the analytical laboratory for PK analysis will be used in all the

analyses. The units of concentration and resulting PK parameters, with amount or concentration in

the unit, will be presented as they are received from the analytical laboratory.

Cmax and tmax will be obtained directly from the plasma concentration-time profiles. For multiple

peaks, the highest post-dose concentration will be reported as Cmax. In the case that multiple peaks

are of equal magnitude, the earliest tmax will be reported.

CCI

Concentrations BLQ from the time of pre-dose sampling (t=0) up to the time of the first quantifiable

concentration will be set to zero with the following exceptions:

• Any embedded BLQ value (between 2 quantifiable concentrations) and BLQ values following

the last quantifiable concentration in a profile will be set to missing for the purposes of PK

analysis.

• If there are late positive concentration values following 2 BLQ concentration values in the

apparent terminal phase, these values will be set to missing, unless there is a scientific

rationale not to do so, which will be documented by the pharmacokineticist.

If an entire concentration-time profile is BLQ, the profile will be excluded from the PK

analysis.

• If a pre-dose concentration is missing, these values may be set to zero by default.

The terminal elimination rate constant ( $\lambda z$ ) will be calculated by log-linear regression of the terminal

portion of the concentration-time profile. The following will be considered:

• If more than one phase is present only data points from the terminal phase will be used.

• A minimum of 3 data points after Cmax, including the last measurable concentration, will be

used for calculating  $\lambda z$ .

• Where the elimination half-life is estimated over less than 3 times the subsequently estimated

terminal half-life the robustness of the  $t\frac{1}{2}\lambda$  estimate will be discussed in the CSR.

• Rsq adjusted should be greater than 0.8. Where Rsq adjusted < 0.8, half-life and half-life

dependent parameters may be excluded from summary statistics and statistical analysis with

sponsor agreement.

The AUCs will be calculated using the linear trapezoidal method when concentrations are increasing

and the logarithmic trapezoidal rule when concentrations are decreasing (linear up log down). The

minimum requirement for the calculation of AUC will be the inclusion of at least 3 consecutive

plasma concentrations above the LLOQ.

Generally, data should not be excluded from analysis. However, where this is scientifically merited a

sensitivity analysis may be performed and the data will be discussed in the CSR.

CCI

Pharmacokinetic summaries will be based upon the PKAS.

Pharmacokinetic parameters will be listed by subject and summarised by treatment. Descriptive statistics for calculated PK parameters will include: n, arithmetic mean, SD, CV%, geometric mean, geometric CV%, median, minimum and maximum values. For tmax, only median, minimum and maximum values will be presented. No descriptive statistics will be determined when fewer than three individual PK parameters are available.

The following rules will be followed with regards to the number of decimal places and presentation of data in the tables and listings for PK parameters:

- Individual PK parameters will be presented to four significant digits, with the exception of tmax, which will be presented to two decimal places.
- Parameters derived directly from source data (e.g. Cmax,) shall be reported with the same precision as the source data (if this is not four significant digits).
- The mean, geometric mean, median and SD values will be reported to four significant digits, all other descriptive statistics will be reported to three significant digits except for CV% which will be presented to one decimal place.
- For tmax the minimum and maximum will be presented to two decimals places and all other descriptive statistics will be presented to three decimal places.

#### 4.13 Other Analyses

Not applicable.

# 4.14 Determination of Sample Size



| I |
|---|

# 4.15 Changes in the Conduct of the Study or Planned Analysis

D6470C00005

The following changes to the statistical methodology planned in Study Protocol will be applied:

• The repeated measures mixed model will also include the time term.

Statistical Analysis Plan

## **5 REFERENCES**

van Genugten RE, van Raalte DH, Muskiet MH, Heymans MW, Pouwels PJW, Ouwens DM, et al. Does dipeptidyl peptidase-4 inhibition prevent the diabetogenic effects of glucocorticoids in men with the metabolic syndrome? A randomised controlled trial. Eur J Endocrinol. 2014 Feb 4;170(3):429-39.

Wan X, Wang W, Liu J, Tong T. Estimating the sample mean and standard deviation from the sample size, median, range and/or interquartile range. BMC Med Res Methodol 2014 Dec 19;14:135.

# 6 APPENDICES

## 6.1 Schedule of Activities

| Visit | 1 | 2 | | | Visi | t 3 a | | | Wash-out | 4 | | | Visi | t 5 a | | | 6 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Phase | Screening | Out-<br>patient<br>visit | Resid | dency | in Un | it <sup>a</sup> | | | (3 weeks) | Out-<br>patient<br>visit | Resid | dency | in Un | it 2 ª | | | Final/ET<br>visit c | Comments |
| Timing | ≤ 14 days<br>before<br>start of | | | | | | | | DAY | | | | | | | | Follow-up<br>30 +/-<br>4 days after | (all sections refer to the<br>CSP) |
| | IMP d | -4 | -2 | -1 | 1 | 2 | 3 | 4 | | 24<br>(-4) | 26<br>(-2) | 27<br>(-1) | 28<br>(1) | 29<br>(2) | 30<br>(3) | 31<br>(4) | last dose of<br>IMP | |
| Informed consent | X | | | | | | | | | | | | | | | | | See Appendix A |
| Verify eligibility criteria | X | | | X | | | | | | | X e | | | | | | | Sections 5.1 and 5.2 |
| COVID-19 symptom telephone screening | X f | X f | X f | | | | | | | X f | X f | | | | | | | Phone call to confirm<br>absence of COVID-19<br>symptoms <sup>f</sup> |
| COVID-19 PCR test | X | | X | | | | | | | | X | | | | | | | Further tests at the discretion of the investigator |
| COVID-19 serology | X | | | | | | | | | | X | | | | | | X | Further tests at the discretion of the investigator |
| Demography | X | | | | | | | | | | | | | | | | | |
| Height and weight | X | | X | | | | | | | | X | | | | | | X | Height at screening only Section 8.3.1 |
| Medical History | X | | | | | | | | | | | | | | | | | |
| Physical examination | X | | Χg | | | | | Χg | | | Χg | | | | | Χg | X | Section 8.3.1 |
| Tobacco use | X | | X | | | | | | | | X | | | | | | | Section 5.3.2 |
| Alcohol breath test | X | | X | | ļ., | | | | | | X | | | | | | | Section 8.3.5.1 |
| Safety ECG | X | | | | X h | | | X | | | | | X h | | | X | X | Section 8.3.3 |
| Vital signs | X | | X | | X h | | | X | | | X | | X h | | | X | X | Section 8.3.2 |
| Randomisation in IVRS | | | X | | | | | | | | | | | | | | | |

CI

| Visit | 1 | 2 | | | Visi | t 3 <sup>a</sup> | | | Wash-out | 4 | | | | t 5 a | | | 6 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Phase | Screening | Out-<br>patient<br>visit | Resid | dency | in Un | it <sup>a</sup> | | | (3 weeks) | Out-<br>patient<br>visit | Resid | dency | in Un | it 2 ª | | | Final/ET<br>visit c | Comments |
| Timing | ≤ 14 days<br>before<br>start of | | | | | | | | DAY | | | | | | | | Follow-up<br>30 +/-<br>4 days after<br>last dose of | (all sections refer to the CSP) |
| | IMP d | -4 | -2 | -1 | 1 | 2 | 3 | 4 | | 24<br>(-4) | 26<br>(-2) | 27<br>(-1) | 28<br>(1) | 29<br>(2) | 30<br>(3) | 31<br>(4) | IMP | |
| Adverse events | | X | X | X | X | X | X | X | | X | X | X | X | X | X | X | X | Section 8.4 |
| Concomitant medication i | X | X | X | X | X | X | X | х | | X | X | X | X | X | X | X | X | Section 6.5 and<br>Appendix F |
| BLOOD SAMPLE COLL | ECTION | | | | • | | | • | | | | | | | | | | • |
| Haematology | X | | X | | X | | | X | | | X | | X | | | X | X | Section 8.3.4 |
| Clinical chemistry<br>(including trigycerides<br>and HDL-C) | Х | | х | | X | | | X | | | X | | X | | | X | х | Section 8.3.4 |
| Coagulation (INR, PT and aPTT) | X | | | | | | | | | | | | | | | | | Section 8.3.4 |
| Serology (HIV I and II,<br>HAV, HbsAg and HCV<br>antibody, tuberculosis) | X | | | | | | | | | | | | | | | | | Section 8.3.4 |
| HbA1c | X | | | | | | | | | | | | | | | | | Section 8.3.4 |
| Pregnancy test (hCG) | X | | | | | | | | | | | | | | | | x | Section 8.3.4. Females only |
| TNFα j | | | | | | | X | | | | | | | | X | | | Pre-dose<br>Post-dose 1, 2, 4, 8, 12,<br>24 hours <sup>k</sup><br>Section 8.2.1.4 |
| PK (AZD9567) | | | | | | | X | х | | | | | | | X | X | | Pre-dose<br>Post-dose<br>5, 0.5, 1, 1.5, 2, 3, 4, 6,<br>8, 12, 24, 30 hours k<br>Section 8.6.1 |

| Visit | 1 | 2 | | | Visi | | | | Wash-out | 4 | | | Visi | | | | 6 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Phase | Screening | Out-<br>patient<br>visit | Resid | dency | in Un | it <sup>a</sup> | | | (3 weeks) | Out-<br>patient<br>visit | Resid | lency | in Uni | t 2 ª | | | Final/ET<br>visit c | Comments |
| Timing | ≤ 14 days<br>before<br>start of | | | | | | | | DAY | | | | | | | | Follow-up<br>30 +/-<br>4 days after<br>last dose of | (all sections refer to the CSP) |
| | IMP d | -4 | -2 | -1 | 1 | 2 | 3 | 4 | | 24<br>(-4) | 26<br>(-2) | 27<br>(-1) | 28<br>(1) | 29<br>(2) | 30<br>(3) | 31<br>(4) | IMP | |
| PK (prednisolone) | | | | | | | X | х | | | | | | | X | X | | Pre-dose<br>Post-dose 0.25, 0.5, 1,<br>1.5, 2, 3, 4, 6, 8, 12, 24,<br>30 hours <sup>k</sup><br>Section 8.6.1 |
| Genetic research | | | X | | | | | | | | | | | | | | | Section 8.8 and<br>Appendix D |
| MMTT | | | | x | | | | х | | | | х | | | | х | | A standardise d mixed meal will be administered around 0700 after an overnight fast. Blood samples to be taken 15 mins preand 10, 20, 30, 60, 75, 120, 180, 240 min post-mixed meal intake (Section 5.3.1) for analysis of plasma glucose, insulin, C-peptide, GLP-1, GIP, glucagon and FFAs, Sections 1.3.1, and 8.2.1.2 |
| Serum cortisol | | | | X | | | X | X | | | | X | | | X | X | X | Sample to be taken at 0800 |

C

| Visit | 1 | 2 | | | Visi | t 3 <sup>a</sup> | | | Wash-out | 4 | | | Visi | t 5 a | | | 6 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Phase | Screening | Out-<br>patient<br>visit | Resid | dency | in Un | it <sup>a</sup> | | | (3 weeks) | Out-<br>patient<br>visit | Resid | dency | in Un | it 2 ª | | | Final/ET<br>visit c | Comments |
| Timing | ≤ 14 days<br>before<br>start of | | | | | | | | DAY | | | | | | | | Follow-up<br>30 +/-<br>4 days after | (all sections refer to the CSP) |
| | IMP d | -4 | -2 | -1 | 1 | 2 | 3 | 4 | | 24<br>(-4) | 26<br>(-2) | 27<br>(-1) | 28<br>(1) | 29<br>(2) | 30<br>(3) | 31<br>(4) | last dose of<br>IMP | |
| CCI | | | | X | | | X | X | | | | X | | | X | X | X | Sample to be taken at 0800 |
| CCI | | | | X | | | X | X | | | | X | | | X | X | X | Sample to be taken at 0800 |
| ACTH | X | | | X | | | X | X | | | | X | | | X | X | X | Fasted sample to be taken at 08:00 |
| CCI | | | | X | | | X | | | | | X | | | X | | | Section 8.2.1.5 |
| URINE SAMPLE COLLE | ECTION | | | | | | | | | | | | | | | | | |
| Urine drug screen<br>(dipstick) | X | | X | | | | | | | | X | | | | | | | Section 8.3.5.1 |
| Urinalysis | X | | X | | X | | | X | | | X | | X | | | X | X | Section 8.3.4 |
| U-Na and U-K | | | | X | | | X | | | | | X | | | X | | | Sampling over 24 h<br>Section 8.2.1.3 |
| Pregnancy test (hCG dipstick) | | | | | X | | | | | | | | X | | | | | Section 8.3.4. Females only |
| STUDY RESIDENCY | | | | | | | | | | | | | | | | | | |
| Admission to CRU | | | X | | | | | | | | X | | | | | | | Admitted to CRU in the<br>early evening on Day -2<br>(approximately 1700) |
| Residency at CRU | | | $\rightarrow$ | | | | | | | | $\rightarrow$ | | | | | | | |
| Discharge from CRU | | | | | | | | X | | | | | | | | X | | Discharge around 1800. |

AL Project Document Version No. Final 2.0
Project Document Effective Date: <Date of last signature>

| Visit | 1 | 2 | | | Visi | t 3 a | | | Wash-out | | | | Vis | it 5 a | | | 6 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Phase | Screening | Out-<br>patient<br>visit | Resid | dency | in Un | it <sup>a</sup> | | | (3 weeks) | Out-<br>patient<br>visit | Resid | dency | in Un | it 2 <sup>a</sup> | | | Final/ET<br>visit c | Comments |
| Timing | ≤ 14 days<br>before<br>start of | | | | | | | | DAY | | | | | | | | Follow-up<br>30 +/-<br>4 days after | (all sections refer to the CSP) |
| | IMP d | -4 | -2 | -1 | 1 | 2 | 3 | 4 | | 24<br>(-4) | 26<br>(-2) | 27<br>(-1) | 28<br>(1) | 29<br>(2) | 30<br>(3) | 31<br>(4) | last dose of<br>IMP | |
| CGM/FGM | | X <sup>1</sup> | X | X | X | X | X | | | X 1 | X | X | X | X | x | | | CGM/FGM will be<br>fitted on an Out-patient'<br>basis on Day -4 and<br>removed on Day 4,<br>Section 8.2.1.1 |
| Standardise d dinner | | | X | | | | X | | | | X | | | | X | | | A standardise d meal<br>will be given at<br>approximately 1900 |
| IMP ADMINISTRATION | | | | | | | | | | | | | | | | | | |
| IMP dosing at clinic | | | | | X | X | X | | | | | | X | X | X | | | Dosing will be around<br>07:00 ( ± 30 min)<br>Section 6 |

- Treatment period 1: Day -4 to Day 4. Treatment period 2: Day 24 to Day 31.
- Wash-out period may be extended to 4 weeks to allow for resolution of acute illness or infection. Further extension needs to be discussed with the investigator.
- Participants who discontinue IMP early (early termination) will have the same assessments as at the Final/ET visit.
- Screening may be extended up to a maximum of 28 days to allow for re-tests to be completed.
- Eligibility criteria to be re-checked before entry to CRU for treatment period 2 (see Section 5.1 and 5.2).
- CRU will call participant 24 hours prior to visit to CRU. Participants should also call the site at any time if they think they may be experiencing COVID-19 symptoms.
- Brief physical examination.
- Pre-dose and 1.5 hours post IMP.
- Participants on dual therapy will require 2 weeks wash-out of SGLT2i or DPP4i.
- TNFα will be measured for high and low dose comparison only (Cohort 1 and Cohort 2).
- PK post-dose timepoints are over two days (ie, reflect one timepoint series).
- CGM/FGM will be fitted on Day -4 to enable 72-hour CGM will be taken at baseline.

# Parexel International

D6470C00005 Statistical Analysis Plan

Note: Interim telephone visits may occur at any time during the Out-patient' periods, as determined by the investigator, to review the safety and well-being of the participant.

Abbreviations: ACTH: adrenocorticotropic hormone; aPTT: activated partial thrombin time; CGM: continuous glucose monitoring; CRU: clinical research unit; DPP4i: Dipeptidyl peptidase-4 inhibitor; ECG: electrocardiogram; ET: end of treatment; FFA: free fatty acid; FGM: flash glucose monitoring; GIP: glucose-dependent insulin releasing polypeptide; GLP-1: glucagon-like peptide-1; HAV: Hepatitis A virus; HbA1c: haemoglobin 1Ac; HbsAg: Hepatitis B surface antigen; hCG: human chorionic gonadotropin; HCV: Hepatitis C virus; HDL-C: High-density lipoprotein-cholesterol; HIV: human immunodeficiency virus; IMP: investigational medicinal product; INR: International normalised ratio; IVRS: Interactive Voice Response System; MMTT: mixed meal tolerance test; PCR: polymerase chain reaction; PK: pharmacokinetics; PT: prothrombin time; SGLT2i: sodium-glucose co-transporter-2 inhibitor; T2DM: type 2 diabetes mellitus; TNFα: tumor necrosis factor alpha; U-K: urinary potassium; U-Na: urinary sodium.

 $\mathbb{CC}$ 

# 6.2 Blood Sampling Schedule for Mixed Meal Tolerance Tests (MMTTs)

| | Day -1, Day 4, Day 27, and Day 31 | Comments |
|---|---|---|
| Plasma glucose, insulin, | 15 10 20 20 (0 55 120 100 210 | |
| C-peptide GLP-1, GIP, | -15, 10, 20, 30, 60, 75, 120, 180, 240 | Time point in relation to the start of the meal |
| glucagon (minutes), and FFAs | | |

GLP-1: glucagon-like peptide-1; GIP: glucose-dependent insulin releasing polypeptide.

CC

# **SIGNATURE PAGE**

This is a representation of an electronic record that was signed electronically and this page is the manifestation of the electronic signature

| Document Name: d6470c00005-sap-ed-3 | | |
|---|---|---|
| <b>Document Title:</b> | Statistical Analysis Plan Edition 3 | |
| Document ID: | CCI | |
| Version Label: | 3.0 CURRENT LATEST APPI | ROVED |
| Server Date<br>(dd-MMM-yyyy HH:mm 'UTC'Z) | Signed by | Meaning of Signature |
| 09-Nov-2021 08:34 UTC | PPD | Quality Assurance Approval |

Notes: (1) Document details as stored in ANGEL, an AstraZeneca document management system.